CLINICAL TRIAL: NCT03236792
Title: Phase 1/2 Study Of Ixazomib In Combination With Cyclophosphamide And Dexamethasone In Patients With Newly Diagnosed Immunoglobulin Light Chain AL Amyloidosis
Brief Title: Ixazomib In Combination With Cyclophosphamide And Dexamethasone for Newly Diagnosed AL Amyloidosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Keren Osman, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-1853
Record Dates: First submitted 2017-07-20; First posted 2017-08-02 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: AL Amyloidosis
Keywords: Newly Diagnosed; AL Amyloidosis; Amyloid; Light chain Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Alzheimer Disease | interventions — ixazomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Newly Diagnosed AL Amyloidosis (Experimental): Ixazomib/Cyclophosphamide/Dexamethasone. Treatment cycles will be repeated up to 6 cycles or until disease progression or until development of significant treatment-related toxicities.
  Interventions: Drug: Ixazomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — 3 mg or 4mg of Ixazomib will be taken orally on days 1, 8, and 15 of a 28-day cycle
Drug: Cyclophosphamide — 300, 400, or 500 mg of oral Cyclophosphamide on days 1, 8, and 15 of a 28-day cycle
Drug: Dexamethasone — 20 mg of oral Dexamethasone on days 1, 8, 15, 22 in a 28-day cycle

SUMMARY:
Light chain (AL) amyloidosis is a bone marrow disorder that affects a wide range of organs that can lead to organ dysfunction and death. Amyloid is an abnormal protein that is produced in your bone marrow and cannot be broken down. It builds up in different organs preventing them from working well. The most commonly affected organs are the kidneys, heart, liver, spleen, nervous system, and digestive tract. Treatment with chemotherapy can stop the growth of abnormal cells that produce this abnormal protein. Decrease in amyloid protein in the body improves the function of the affected organs.

The primary purpose of this study is to determine the safest dose of the medications and how well you tolerate them or the "maximum tolerated dose" (MTD). The study uses Ixazomib in combination with cyclophosphamide and dexamethasone to treat people with newly diagnosed AL amyloidosis. This combination of medications is an oral regimen that is taken over 6 cycles. The first part of study will determine the safety of this regimen and the second part of the study will determine how effective this combination of drugs is to treat your disease.

DETAILED DESCRIPTION:
This study is a phase 1/2 study to assess safety and hematologic response rate of Ixazomib (MLN) in combination with Cyclophosphamide (CTX) and Dexamethasone (DEX). This is an open label multi-center, dose escalation safety study for patients with newly diagnosed AL Amyloidosis.

A 3+3 design will be utilized to determine the MTD for MLN + CTX + DEX in 28-day treatment cycle. Treatment cycles will be repeated up to 6 cycles or until disease progression or until development of significant treatment-related toxicities. A total of up to 30 patients are planned to enroll into the study, with a maximum of 18 patients in the dose escalation arm and 18 patients in the MTD expansion arm. The cohort of 6 patients treated at the MTD during the dose expansion phase will also serve as the initial 6 patients for the expansion Phase II cohort. These 6 patients will contribute data to both the phase I dose escalation study and the phase II expansion study. To complete the Phase II cohort, an additional 12 new patients will need to be enrolled.

MLN will be taken orally on days 1, 8, and 15 at doses of 3 mg or 4 mg. CTX will be taken orally on the same days with dose escalation from 300 mg up to 500 mg. DEX will be taken orally on days 1, 8, 15, 22 at 20 mg in the 28-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older.
* Biopsy-proven diagnosis of AL amyloidosis according to the following standard criteria:

  * Histochemical diagnosis of amyloidosis, as based on tissue specimens with Congo red staining with exhibition of an apple-green birefringence
  * If clinical and laboratory parameters insufficient to establish AL amyloidosis or in cases of doubt, amyloid typing may be necessary
  * Measurable disease defined by serum differential free light chain concentration (difference between amyloid forming [involved] and non amyloid forming [uninvolved] free light chain [FLC]) ≥ 50 mg/L).
  * Amyloid organ involvement including renal, cardiac, GI and/or nervous system involvement as well as soft tissue disease
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2.
* Patients must meet the following clinical laboratory criteria:

  * Absolute neutrophil count (ANC) ≥1,000/mm3 and platelet count ≥75,000/mm3.
  * Hemoglobin ≥ 8.0 g/dL
  * Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
  * Total bilirubin ≤ 2 the upper limit of the normal range (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 x ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 ULN.
  * Calculated creatinine clearance ≥ 30 mL/min (Cockcroft-Gault Formula).

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Major surgery within 14 days before enrollment.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
* Evidence of current uncontrolled cardiovascular conditions:

  * uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, *unstable angina, or myocardial infarction within the past 6 months.

Recent history of myocardial infarction in the six months prior to registration

* Systemic treatment, within 14 days before the first dose of ixazomib, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with early stage prostate cancer, non melanoma skin cancer or carcinoma in situ of any type are not excluded; patients with malignancies that have undergone complete resection are not excluded.
* Patient has ≥ Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 21days of the start of this trial and throughout the duration of this trial.
* New York Heart Association Class III or IV Heart Failure
* NT Pro-BNP > 8500pcg/mL.
* Dialysis dependent renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | up to 3 years
  The MTD of ixazomib given in combination with cyclophosphamide and dexamethasone, 3 + 3 design in Phase 1 of this study

SECONDARY OUTCOMES:
Response Rate | up to 3 years
  The incidence of hematologic response rate as defined by complete response (CR), very good partial response (VGPR), partial response (PR), and stable disease (SD)
Frequency of organ response | up to 3 years
  The frequency of organ response as per the ISA criteria: Cardiac response and progression -NT-proBNP response (>30% and > 300 ng/L decrease if baseline NT-proBNP 650 ng/L). NT-proBNP progression (>30% and >300 ng/L increase). cTn progression (>33% increase). NYHA class response (> two-class decrease if baseline NYHA class 3 or 4). EF progression (>10% decrease). Renal response and progression - Renal response: >30% decrease in proteinuria or drop of proteinuria below 0.5 g/24 h in the absence of renal progression. Renal progression: >25% decrease in eGFR. Liver response criteria- include a 50% decrease in abnormal alkaline phosphatase value and decrease in liver size of at least 2cm.

CONTACTS AND LOCATIONS:
Overall Officials: Keren Osman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided